CLINICAL TRIAL: NCT02810093
Title: SENOMETRY : Big Data and Text-mining Technologies Applied for Breast Cancer Medical Data Analysis
Brief Title: Big Data and Text-mining Technologies Applied for Breast Cancer Medical Data Analysis
Acronym: SENOMETRY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Quantmetry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 6373
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Text mining; Big Data; Machine Learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients between 2000 and 2016: Patients treated for a breast cancer between 2000 and 2016 in the Hospital of Strasbourg (France).
  Interventions: Other: retrospective medical records analyze

INTERVENTIONS:
Other: retrospective medical records analyze — Ten thousand medical records (between years 2000 and 2016) will be analyzed

SUMMARY:
Primary purpose :

To develop a method to automatically extract and structure the information included in numerous medical records from breast cancer patients.

Secondary purpose :

With this procedure we can analyze the content of ten thousand anonymized textual medical records.

This information should enable us to explore many subjects, such as:

* The impact of certain therapeutic procedures
* The characteristics of sub-groups of patients
* Pregnancy associated breast cancers
* Risk factors

ELIGIBILITY:
Inclusion Criteria:

* Majority (age > 18)
* Malignant breast tumors
* signed informed consent

Exclusion Criteria:

* Benign breast pathology
* Patients not initially treated at the Hôpitaux Universitaires de Strasbourg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (men and women) suffering from an in situ or invasive cancer treated at Hôpitaux Universitaires de Strasbourg between years 2000 and 2016.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Validate the reliability of a computer-based, automatic information retrieval method specific to medical records from breast cancer multidisciplinary meetings | 6 months

SECONDARY OUTCOMES:
Breast cancer recurrence rate after some therapeutic procedures | 6 months
  Study of the recurrence rate of different subgroups of patients where various procedures were performed

CONTACTS AND LOCATIONS:
Overall Officials: Carole Mathelin, MD, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- University Strasbourg Hospital, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simoulin A, Thiebaut N, Neuberger K, Ibnouhsein I, Brunel N, Vine R, Bousquet N, Latapy J, Reix N, Moliere S, Lodi M, Mathelin C. From free-text electronic health records to structured cohorts: Onconum, an innovative methodology for real-world data mining in breast cancer. Comput Methods Programs Biomed. 2023 Oct;240:107693. doi: 10.1016/j.cmpb.2023.107693. Epub 2023 Jun 25. PMID 37453367